CLINICAL TRIAL: NCT03220880
Title: Clinical Characteristics of Intranasal Dexmedetomidine for Sedation in Children Undergoing Non-painful Procedures
Brief Title: Intranasal Dexmedetomidine Sedation in Children for Non-painful Procedures
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Children's Healthcare of Atlanta (Other); University of Pittsburgh (Other); Children's Hospital Medical Center, Cincinnati (Other); UNC Children's Hospital (Unknown); Santa Clara Valley Medical Center (Other); Baylor College of Medicine (Other); HSHS St. John's Hospital (Unknown); Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Daniel S Tsze, MD, MPH, Associate Professor of Pediatrics in Emergency Medicine at CUMC, Columbia University
Other Study IDs: AAAR5010
Record Dates: First submitted 2017-07-14; First posted 2017-07-18 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Dexmedetomidine; Sedation
Keywords: Dexmedetomidine; Sedation; Pediatric

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Intranasal dexmedetomidine: Intranasal dexmedetomidine (100 mcg/mL), 0.5 to 4 mcg/kg
  Interventions: Drug: Intranasal dexmedetomidine

INTERVENTIONS:
Drug: Intranasal dexmedetomidine — Intranasal dexemedetomidine (100 mcg/mL), 0.5 to 4 mcg/kg

SUMMARY:
Specific Aim 1: To describe the adequacy of sedation associated with different regimens of IN DEX in children undergoing non-painful procedures. This aim will test the working hypothesis that IN DEX regimens are effective for producing sedation adequate for completion of non-painful procedures in children.

Specific Aim 2: To describe the temporal characteristics associated with varied regimens of IN DEX in children undergoing non-painful procedures, such as time to onset of adequate sedation; time to procedure start; and time from procedure end to meeting discharge criteria. This aim will test the working hypothesis that IN DEX regimens have temporal characteristics that are favourable for sedating children for non-painful procedures.

Specific Aim 3: To describe the adverse events associated with varied regimens of IN DEX in children undergoing non-painful procedures. This aim will test the working hypothesis that IN DEX regimens have a low incidence of adverse events.

DETAILED DESCRIPTION:
Dexmedetomidine (DEX) is an alpha-2 receptor agonist with sedative, anxiolytic, and analgesics properties. DEX has been used extensively for sedation in children to facilitate different non-painful procedures, such magnetic resonance imaging (MRI), auditory brainstem response (ABR) tests, and computed tomography (CT) scans. In particular, DEX can be administered by the intranasal (IN) route. Intranasal administration has the benefits of being both effective and needle-free, of which the latter makes it less distressing to children compared to sedatives administered by the intravenous (IV) route. There is a gap of knowledge, however, regarding the ideal regimen of IN DEX for providing optimal procedural sedation in children undergoing non-painful procedures. There is a large variation in practice using IN DEX, both regarding the dose and the use of adjunct medications. It is also unknown whether regimens should vary based on patient factors such as age. There is no clear evidence to define best practice when using IN DEX to provide sedation in this population to achieve the desired outcomes most relevant to clinicians. The rationale of the proposed investigation is that by conducting an exploratory study to measure clinical outcomes associated with IN DEX, the investigators can begin to identify trends and differences that will lay the foundation for randomized clinical trials to identify the ideal regimen for IN DEX when providing sedation for non-painful procedures. This will then allow the investigators to compare IN DEX, at its best, to other sedatives so that the sedative and regimen associated with the best outcomes relevant to sedation of children undergoing non-painful procedures can be determined.

ELIGIBILITY:
Inclusion Criteria:

* Children 2 months to 17 years (i.e. before their 18th birthday)
* Child will be receiving intranasal dexmedetomidine as part of their usual medical care
* Child will be undergoing a non-painful medical procedure, which includes (but is not limited to): MRI, CT scans, ABR/BAER, echocardiograms, and EEGs.

Exclusion Criteria:

* Known allergy to dexmedetomidine
* Known abnormal renal or hepatic function
* Known cardiac conduction abnormality or heart block
* Current use of digoxin or beta-blockers

Ages: 2 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children undergoing sedation using intranasal dexmedetomidine for non-painful procedures.
Sampling Method: Non-Probability Sample
Enrollment: 578 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Adequacy of sedation | 1 hour
  Pediatric Sedation State Scale

SECONDARY OUTCOMES:
Time to onset of adequate sedation | 1 hour
  Time in minutes after administration of IN DEX to achieve a University of Michigan Sedation Scale (UMSS) score of 3 or more
Time to discharge | 2 hours
  Time in minutes after procedure end to achieving Modified Aldrete Scoring System (MASS) score of 9 or greater, or baseline MASS score.

OTHER OUTCOMES:
Adverse events | 3 hours
  Adverse events and/or required interventions (e.g. cardiovascular, airway) required

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Tsze, MD, MPH, Principal Investigator — Columbia University
Locations (8):
- United States (8):
  - Santa Clara Valley Medical Center, San Jose, California
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Southern Illinois University Healthcare, Springfield, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - UNC Children's Hospital, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

REFERENCES:
- [Derived] Tsze DS, Rogers AP, Baier NM, Paquin JR, Majcina R, Phelps JR, Hollenbeck A, Sulton CD, Cravero JP. Clinical Outcomes Associated With Intranasal Dexmedetomidine Sedation in Children. Hosp Pediatr. 2023 Mar 1;13(3):223-243. doi: 10.1542/hpeds.2022-007007. PMID 36810939